CLINICAL TRIAL: NCT03834779
Title: A Community-Clinic Collaboration to Improve Outcomes in HIV+ Substance Users Released From Jail
Brief Title: HIV+ Substance Users Released From Jail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ank Nijhawan, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU 082017-022; 1R34DA045592-01 (NIH)
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: HIV/AIDS; Substance Use Disorders
Keywords: HIV; AIDS; Substance Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOORS-CHW Intervention (Other): The type of intervention is behavioral.
  Participants randomized to the intervention arm will meet with the Community Health Worker (CHW) and a staff member from Unlocking DOORS. The Unlocking DOORS broker will complete a needs assessment, generate an individualized re-entry plan and make referrals to providers in the extensive Unlocking DOORS network. The CHW will assist the participant in navigating these referrals, specifically with regards to HIV care, substance use treatment and mental healthcare.
  Interventions: Behavioral: DOORS-CHW Intervention
- Treatment As Usual (No Intervention): TAU participants will receive standard of care, which involves passive referral by jail medical staff to the outpatient HIV clinic.

INTERVENTIONS:
Behavioral: DOORS-CHW Intervention — The behavioral intervention has been developed for a collaborative CHW and re-entry program intervention that targets HIV outcomes, substance use and recidivism in HIV+ jail releasees.
  Participants will be randomized to the DOORS+CHW intervention versus TAU and all participants will undergo study follow-up visits at 3, 6 and 12 months. In other words, participants randomized to the intervention arm will meet with the CHW and a staff member from DOORS. One of the primary study aims is a randomized controlled trial of an intervention which has a reasonable probability of improving the health and well-being of the subject by improving linkage to social services and the HIV clinic. The control arm will receive standard of care (referrals to case management).
  Arms: DOORS-CHW Intervention

SUMMARY:
The long-term goal of this project is to improve HIV and substance use outcomes and reduce recidivism for HIV+ substance users released from jail. The overall objective of the proposed R34 project is to develop and pilot test a multi-sector community-clinic collaborative intervention that can subsequently be implemented on a larger scale (as part of a future R01) to achieve this goal. Our central hypothesis is that HIV+ substance users released from jail can successfully overcome obstacles to re-entry and continuity of HIV care with individualized, culturally competent assistance in navigating both social and medical services.

Aim 1: Develop and refine a collaborative CHW and re-entry program intervention that targets HIV outcomes, substance use and recidivism in HIV+ jail releasees.

Aim 2: Conduct a pilot randomized controlled trial comparing the collaborative intervention (n=40) compared to treatment as usual (n=40) in HIV+ substance users released from jail.

DETAILED DESCRIPTION:
Aim 1 Introduction: This first aim will be critical to successful implementation of the CHW-DOORS intervention. Employing a formerly incarcerated CHW to assist individuals leaving prison in order to connect to healthcare has been successfully implemented in different settings, but it has not been applied specifically to HIV patients or those leaving jail (v. prison), nor has it been integrated into a community based organization. The objective of this aim is to adapt the evidence-based CHW intervention to the HIV population and to the jail setting and to integrate the CHW into existing processes at DOORS and the outpatient HIV clinic system.

Research Design. Aim 1.1: The first step of Aim 1 will be to train the CHW using the transitions clinic approach, add modules on HIV and substance use and familiarize the CHW with DOORS processes and HIV clinic workflow.

Aim 1.2: The second step will be to complete qualitative interviews with stakeholders in three different settings- the jail, the HIV clinic and DOORS. All interviews will be semi-structured, one-on-one interviews, with an estimated 4-7 interviews in each setting.

The structured component of the interview guide will prompt interviewee input on study design (e.g. recruitment, intervention, follow-up visits), content of the intervention (e.g. high demand services) and an open-ended component eliciting possible barriers to study implementation.

Aim 1.3: The final step in Aim 1 will be to complete pilot testing with 5 subjects, which will focus on refining recruitment/enrollment protocols, streamlining study assessments and evaluating the intervention.

Recruitment: In order to protect patient confidentiality, potential subjects will be referred by medical staff who provide clinical care to HIV+ inmates. When an inmate enters the Dallas County Jail, he/she is evaluated by a medical provider within 24 hours (medical assessment program, MAP). At this visit, the inmate can disclose any medical conditions that they have including HIV, in which case he/she will be referred to the jail HIV clinic (scheduled within 1-7 days of jail entry). In addition, HIV testing is offered in an opt-out manner when inmates have blood drawn for any reason (approximately 10% of jail population) and by inmate request, and those with positive test results are referred to jail HIV clinic. Candidates coming through the MAP or HIV clinics who agree to be approached will be contacted by a research assistant (RA). The RA will explain the study to interested individuals, will obtain additional contact information (additional phone numbers, address or location in community where patient could be found) and permission to contact the individual after release. Clinic staff will also routinely request this information from interested individuals in case they are released prior to RA visit in jail. Once released, the research team will contact the individual releasee to schedule an enrollment visit. At this visit, which will occur as soon as possible after jail release (maximum within 30 days of release), the research team will obtain informed consent and enroll the participant into the study. The enrollment may occur at the UT Southwestern HIV research unit (located above the main HIV clinic) or in the community as per participant preference.

Enrollment: In order to be enrolled, individuals must (a) be ≥18 years old, (b) have a confirmed diagnosis of HIV, (c) have evidence of uncontrolled HIV (viral load >200 copies/mL within 90 days of enrollment, self-reported non-adherence to HIV medications or no community clinic visit in the 6 months preceding incarceration), (d) report or have medical records documenting any opioid (illicit or prescription misuse), stimulant (cocaine, ecstasy, or amphetamines), or heavy alcohol use (as determined by the 3-item Alcohol Use Disorders Identification Test (AUDIT-C) within the past 12 months, and (e) provide at least 2 forms of contact information. They will also be asked to provide a release of information for their medical records at the jail and community clinics/ hospitals. No randomization will occur in Aim 1 as all 5 participants in the pilot testing phase will be assigned to the intervention. Baseline assessments will occur after informed consent is obtained and enrollment is complete. These assessments will focus on variables in the conceptual model, with collection of demographics (age, race/ethnicity, gender, HIV risk factor) and social variables (marital status, housing, education, employment/income, insurance, benefits, social support). Subjects will also be asked about HIV care (engagement in care, antiretroviral therapy, adherence to medications (using visual analog scale), barriers to care), mental illness, and substance use (using ASSIST questionnaire).

Intervention: The first meeting with the CHW will occur at the time of enrollment if possible, depending on availability of the participant and CHW, otherwise it may occur anytime within 14 days of enrollment. After release from jail, the CHW will help the participant navigate to DOORS, where they will meet with a "broker", someone who helps the client/participant arrange and negotiate referrals to services within the extensive partner/provider network. The first broker meeting will typically occur within 2-4 weeks after release, as this is a critical window for re-engagement in care, underscored by the fact that this is also a high-risk period for increased unprotected sex and return to substance use. Per DOORS' standard practice, the broker will complete a comprehensive needs assessment with the participant. Based on these assessments, together with the participant, the broker will develop a personalized re-entry plan with a detailed list of referrals and calendar of scheduled visits with relevant agencies within the DOORS network.

Follow-up visits and assessments: Research visits will be scheduled at 3 months, 6 months and 12 months. A 4-week window before and 8-week window after the target follow-up dates will be permitted for study assessments. Assessments will be completed at each follow-up visit, including substance use, adherence, healthcare utilization and recidivism, with blood draw for HIV viral load collected at the 6-month visit. In order to maximize efficient utilization of resources, for baseline and other follow-up visits, HIV viral load will be abstracted from medical records. In order to have sufficient time to enroll and complete 12 month study visits for the 80 participants in Aim 2, the 5 pilot participants from Aim 1.3 need to reach at least the 3 month time point but not 6 or 12-month visits before beginning study enrollment for Aim 2. Pilot participants will complete through 12-month visits as this will provide insight as to how best to conduct these later follow-up visits. All participants will receive financial reimbursement for study visits ($25 for each visit), unless they are incarcerated at the time of the visit. Jail inmates are not permitted to receive any financial incentives during incarceration.

AIM 2: Conduct a pilot randomized controlled trial comparing the collaborative intervention (n=40) compared to treatment as usual (n=40) in HIV+ substance users released from jail.

Introduction. In this aim, we will test the CHW-DOORS intervention that was refined in Aim 1 in a randomized fashion. The goal of this aim is to establish feasibility of a randomized controlled trial in this setting, to determine preliminary efficacy of the intervention and to inform sample size calculations for a fully powered trial. In addition, this aim will provide data regarding key factors involved in HIV+ substance users accessing substance use treatment and HIV care after jail release. Our working hypothesis is that from the stakeholder input and pilot testing completed in Aim 1, we will be able to successfully conduct a pilot randomized controlled trial and gain valuable insight into key predisposing and enabling factors influencing healthcare needs and utilization in this population, and how these may impact HIV viral load, substance use and recidivism.

Research Design. Potential participants will be referred to the research study by Dallas County jail medical providers as described in Aim 1.3. Candidates who agree to be approached will be contacted by a RA who will recruit, and review eligibility criteria (see Aim 1.3). After release, potential participants will be contacted in order to complete informed consent, study enrollment and randomization (to be completed within 30 days of release from jail). All participants will provide 2 specific forms of locator information (telephone number for themselves, friend/family member, address, email, specific location where they may be located to aid in retention efforts). Participants will complete baseline assessments and will then be randomized to the intervention CHW-DOORS versus treatment as usual (TAU). Randomization will occur by random assignment using a computer program, without block randomization given the small sample size. TAU participants will receive standard of care, which involves passive referral by jail medical staff to the outpatient HIV clinic.

Intervention. Participants randomized to the intervention arm will meet with the CHW and a staff member from DOORS as outlined in Aim 1.3. Any modifications to this protocol after pilot testing in Aim 1.3 will be implemented in Aim 2. The general premise will be the same, where the DOORS broker will complete a needs assessment, generate an individualized re-entry plan and make referrals to providers in the extensive DOORS network. The CHW will assist the participant in navigating these referrals, specifically with regards to HIV care, substance use treatment and mental healthcare. The measurement of the intervention will be as noted in Aim 1.3, with the DOORS broker following routine agency processes for referrals and measurement using the PIECES technology program and the CHW will record specifics (where, when, duration) of each visit and what was addressed during these intervention visits.

Study Assessments. All participants will complete baseline assessments prior to randomization and will have follow-up visits at 3, 6 and 12 months as noted in Aim 1.3. A blood draw will be performed for 6-month HIV viral load. Follow-up visits will assess HIV viral load (abstracted from medical record for all visits other than 6 month), substance use (using ASSIST), healthcare utilization including attendance of HIV clinic visits, emergency room visits, hospitalizations and reincarceration. If individuals are reincarcerated at the Dallas County Jail at the time of the follow-up visits, an attempt will be made to complete study visits at the jail.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected AND
* ≥18 years old AND
* report or have medical records documenting any opioid (illicit or prescription misuse), stimulant (cocaine, ecstasy, or amphetamines), or heavy alcohol use (as determined by the 3-item Alcohol Use Disorders Identification Test (AUDIT-C) within the past 12 months
* Provide two forms of contact information (address, phone number, email, other locator info) AND
* HIV VL >200 copies/mL within past 90 days OR
* No HIV visit in 6 months OR Self-reported non-adherence to medications

Exclusion Criteria:

* Unwilling to participate
* Unable to consent
* Does not speak English
* Unwilling to participate
* Unable to consent
* Does not plan to remain in greater Dallas area after release Sentenced to prison or other court-mandated program for ≥6 months
* Does not speak English
* Have an acute medical or psychiatric disorder that would, in the judgment of the PI, make participation difficult or unsafe.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ank E Nijhawan, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Amelia Court, HIV Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study and there was not direct mention of data sharing in the informed consent form, there is not plan to share IPD with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 individuals enrolled and assigned to study arms, all 31 who were enrolled were deemed eligible
Groups:
- DOORS-CHW Intervention: The type of intervention is behavioral.
  Participants randomized to the intervention arm will meet with the Community Health Worker (CHW) and a staff member from Unlocking DOORS. The Unlocking DOORS broker will complete a needs assessment, generate an individualized re-entry plan and make referrals to providers in the extensive Unlocking DOORS network. The CHW will assist the participant in navigating these referrals, specifically with regards to HIV care, substance use treatment and mental healthcare.
  DOORS-CHW Intervention: The behavioral intervention has been developed for a collaborative CHW and re-entry program intervention that targets HIV outcomes, substance use and recidivism in HIV+ jail releasees.
  Participants will be randomized to the DOORS+CHW intervention versus TAU and all participants will undergo study follow-up visits at 3, 6 and 12 months.
Period: Overall Study
Arm/Group | DOORS-CHW Intervention | Treatment As Usual
Started | 17 | 14
Completed | 10 | 8
Not Completed | 7 | 6
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Population: Analysis population same as assigned treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | DOORS-CHW Intervention | Treatment As Usual | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (9.7) | 34.7 (9.3) | 35.9 (9.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 12 | 12 | 24
  Gender: Female | 3 | 1 | 4
  Gender: Transgender female | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 2 | 3 | 5
  Race/ethnicity: Non-Hispanic Black | 13 | 9 | 22
  Race/ethnicity: Hispanic | 2 | 2 | 4
CD count [Mean (Standard Deviation); unit: cells per cubic millimeter of blood] — CD4 count is measured at baseline as cells per cubic millimeter of blood
  cells per cubic millimeter of blood | 412 (359) | 371 (275) | 388 (306)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable HIV Viral Load
Description: Number of participants with an undetectable HIV viral load (<200 copies/mL) is assessed via blood work.
Time Frame: At 6 months after enrollment
Population: All participants who had viral load completed at 6 months
Measure: Count of Participants; unit: Participants
Groups:
- DOORS-CHW Intervention: The type of intervention is behavioral.
  Participants randomized to the intervention arm will meet with the Community Health Worker (CHW) and a staff member from Unlocking DOORS. The Unlocking DOORS broker will complete a needs assessment, generate an individualized re-entry plan and make referrals to providers in the extensive Unlocking DOORS network. The CHW will assist the participant in navigating these referrals, specifically with regards to HIV care, substance use treatment and mental healthcare.
  DOORS-CHW Intervention: The behavioral intervention has been developed for a collaborative CHW and re-entry program intervention that targets HIV outcomes, substance use and recidivism in HIV+ jail releasees.
  Participants will be randomized to the DOORS+CHW intervention versus TAU and all participants will undergo study follow-up visits at 3, 6 and 12 months. In other words, participants randomized to the intervention arm will meet with the CHW and a staff member from DOORS. One of the primary study aims is a randomized controlled trial of an intervention which has a reasonable probability of improving the health and well-being of the subject by improving linkage to social services and the HIV clinic. The control arm will receive standard of care (referrals to case management).
Arm/Group | DOORS-CHW Intervention | Treatment As Usual
Number analyzed (Participants) | 10 | 8
Participants | 2 | 3

2. Secondary Outcome: Number of Participants Who Are Positive/Negative for Substance Use as Assessed Via Urine Drug Screen
Description: Number of participants who are positive/negative for Substance use are assessed via urine drug screen
Time Frame: At 6 months after enrollment
Population: All participants who had urine toxicology screen at 6 months were assessed
Measure: Count of Participants; unit: Participants
Arm/Group | DOORS-CHW Intervention | Treatment As Usual
Number analyzed (Participants) | 9 | 9
Participants
  positive for stimulants | 4 | 8
  not positive for stimulants | 5 | 1

3. Other Pre Specified Outcome: Change in Substance Use for Reported Drug of Choice From Baseline at 6 Months After Enrollment as Assessed Via ASSIST Questionnaire
Description: Change in substance use from baseline at 6 months after enrollment (result reported is the baseline minus the 6 month value) is assessed via ASSIST(Alcohol, Smoking, and Substance Involvement Screening Test) v3.1 questionnaire. For the participant's reported DRUG OF CHOICE, the score on the relevant subscale will be used: (A) ASSIST risk score for tobacco (range 0-31); (B) alcohol (range 0-39); (C) cannabis (range 0-39); (D) cocaine (range 0-39); (E) amphetamine-type stimulants (range 0-39); (F) inhalants (range 0-39); (G) for sedatives or sleeping pills (range 0-39); (H) hallucinogens (range 0-39); (I) opioids (range 0-39); (J) 'other' drugs (range 0-39); High values indicate a worse outcome. Subscales are not combined;
  Score interpretation:
  Lower Risk: Alcohol (0-10), All other substances (0-3); Moderate Risk: Alcohol (11-26), All other substances (4-26); High risk: Alcohol (26+), All other substances (27+);
Time Frame: Baseline and 6 months after enrollment
Population: participants completing ASSIST score at baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DOORS-CHW Intervention | Treatment As Usual
Number analyzed (Participants) | 13 | 11
score on a scale
  All | 5.7 (14.9) | 12 (12.8)
  Participants with tobacco as their drug of choice: number analyzed (Participants) | 0 | 0
  Participants with alcohol as their drug of choice: number analyzed (Participants) | 1 | 1
  Participants with alcohol as their drug of choice | 10 (0) | -3 (0)
  Participants with cannabis as their drug of choice: number analyzed (Participants) | 0 | 0
  Participants with cocaine as their drug of choice: number analyzed (Participants) | 6 | 5
  Participants with cocaine as their drug of choice | -16.2 (16.7) | -4.8 (8.7)
  Participants with amphetamine-type stimulants as their drug of choice: number analyzed (Participants) | 4 | 5
  Participants with amphetamine-type stimulants as their drug of choice | -14.3 (11.8) | -1.6 (7.9)
  Participants with inhalants as their drug of choice: number analyzed (Participants) | 0 | 0
  Participants with sedatives or sleeping pills as their drug of choice: number analyzed (Participants) | 0 | 0
  Participants with hallucinogens as their drug of choice: number analyzed (Participants) | 1 | 0
  Participants with hallucinogens as their drug of choice | -24 (0) |
  Participants with opioids as their drug of choice: number analyzed (Participants) | 1 | 0
  Participants with opioids as their drug of choice | -3 (0) |
  Participants with 'other' drugs as their drug of choice: number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Number of Participants Who Experienced Recidivism
Description: Number of participants who experienced recidivism is measured by the count of participants who had a re-incarceration in jail or prison at 12 months
Time Frame: at 12 months after enrollment
Population: participants who were alive at the end of the study and were reincarcerated
Measure: Number; unit: participants
Arm/Group | DOORS-CHW Intervention | Treatment As Usual
Number analyzed (Participants) | 16 | 12
participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | DOORS-CHW Intervention | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 1/17 | 2/14
Serious Adverse Events (participants affected / at risk) | 12/17 | 6/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOORS-CHW Intervention (N=17) | Treatment As Usual (N=14)
Hospitalization (General disorders) | 12 (12) | 6 (6) — Inpatient stay

LIMITATIONS AND CAVEATS:
Limitations: This study (1) was initiated just before the COVID-19 pandemic which limited recruitment and decreased opportunities for in-person interaction between participants and staff. However, efforts were made to connect with participants outdoors or through virtual methods whenever possible. (2) is a single center study localized in a large Southern city with a focus on both substance use - primarily stimulants - and HIV and therefore may not be applicable to other locations/populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03834779/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03834779/SAP_001.pdf
  • Informed Consent Form (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03834779/ICF_002.pdf